CLINICAL TRIAL: NCT06543641
Title: Evaluation of Long Coronary Artery Stents With Third-generation Dual-source Computed Tomography Angiography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lauri Mansikkaniemi (Other)
Responsible Party: Sponsor-Investigator, Lauri Mansikkaniemi, M.D., Helsinki University Central Hospital
Organization: Helsinki University Central Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: M1016TUTLA
Record Dates: First submitted 2024-07-25; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Coronary Artery Disease; Chronic Total Occlusion of Coronary Artery
Keywords: coronary artery disease; drug-eluting stent; percutaneous coronary intervention; coronary computed tomography angiography
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Masking Description: The study's cardiac radiologist was blinded for symptomatic data, stent type and stent quantity. The target vessel of implanted coronary artery stents was provided.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study population (Other): All patients included in the study.
  Interventions: Diagnostic Test: Coronary computed tomography angiography; Diagnostic Test: Invasive coronary angiography

INTERVENTIONS:
Diagnostic Test: Coronary computed tomography angiography — All patients received coronary computed tomography angiography.
  Other Names: CCTA
Diagnostic Test: Invasive coronary angiography — According to the study criteria some of the patients received confirmation imaging with invasive coronary angiography.
  Other Names: ICA

SUMMARY:
The goal of this clinical trial is to assess third-generation dual-source coronary computed tomography angiography (CCTA) performance in the evaluation of long coronary stents in patients with coronary artery chronic total occlusions. The main questions it aims to answer are:

* Can patency of long coronary artery stents be assessed with third generation CCTA?
* What are the factors affecting the assessability?
* What is the radiation exposure of third generation CCTA?

DETAILED DESCRIPTION:
This prospective study complied with the Declaration of Helsinki and was approved by the ethics committee of Helsinki University Central Hospital. All patients gave a written informed consent prior to the beginning of the study.

Patient selection A registry that included chronic total occlusion (CTO) patients with stable coronary artery disease treated for CTO with percutaneous coronary angioplasty (CTO PCI) in Helsinki University Central Hospital starting from 2014 was used for this study. The study population included consecutive, prospectively recruited patients from 2014 to 2019. All patients meeting the study criteria were included in the study.

Definition Segments 5 mm proximal and 5 mm distal to the stent were considered as part of the stent for in-stent restenosis (ISR) evaluation, as proposed by the Academic Research Consortium and were included in CCTA performance analyses. Long CTO stents consisted of one or more coronary artery stents with possible combination of different stent types. The combined stent length was reported without possible overlap for multiple stents. The diameter of the largest stent or post-dilation balloon was reported. Based on previous CT studies and guidelines radiological ISR in CCTA was defined as luminal narrowing of ≥ 50% in the long CTO stent. CCTA result was considered negative if ISR was ruled out and positive if ISR was detected or if the result was inconclusive. Therefore, two groups defined by the CCTA result were formed. In patient-based analyses patients with two long CTO stents of which at least one was a CCTA positive stent were considered as CCTA positive. In native coronary arteries less than 25% was considered minimal, 25-49% mild, 50-69% moderate and 70-99% severe stenosis and 100% as an occlusion. Assessment of stenosis was based on direct visualisation. The study's experienced cardiac radiologist with over 15 years of experience was blinded for symptomatic data, stent type and stent quantity. The target vessel of implanted coronary artery stents was provided.

All patients underwent third-generation dual-source CCTA. In CCTA a non-contrast calcium score using standard 120 kilovolt (kV) acquisition and 3 mm slice thickness was obtained. Stented segments were manually subtracted from the score. Second, third-generation dual-source CCTA (Somatom Force, Siemens) was performed. Prospective ECG-triggering was applied regular heart rate < 70/min and/or in the case of previous stent implantation of right coronary artery (RCA) to avoid motion artefacts and FLASH- mode if the heart rate was regular and < 60/min. If the presenting heart rate was > 70/min, metoprolol 5-15 mg was administered intravenously. For patients with higher heart rates (> 70/min) prospective ECG-gating and widening of the acquisition window (padding) were used. Sublingual nitroglycerin was administered before scanning. A tube voltage of 100 kV, rotation time of 0.25 s, temporal resolution of 66 ms, collimation of 2 x 192 x 0.6 mm and pitch of 3.2 were used. Approximately 50 ml of contrast medium containing 350 mg/ml of iodine (Omnipaque 350, GE Healthcare) was injected intravenously at a flow rate of 5-5.7 ml/s, followed by a 47 ml saline solute. Axial images were reconstructed with 0.6 mm slice and evaluated using multiplanar reformation. Bv40 kernel, Advanced Modeled Iterative Reconstruction 3 (ADMIRE 3) and Iterative metal artefact reduction (iMAR) were utilised.

Clinical information and CCTA results were assessed by the interventional cardiologists and the following patients were offered invasive coronary angiography (ICA):

1. Patients with a positive result in a long CTO stent
2. Patients with a positive result in a non-CTO stent
3. Patients with ≥ 50% stenosis or an inconclusive finding in any native coronary artery in patients with anginal symptoms.

Physiological evaluation (fractional flow reserve) and intravascular imaging (intravascular ultrasound, optical coherence tomography) were performed in ICA by the decision of the interventional cardiologist. Any incidental findings were evaluated separately.

Radiation exposures of CCTA and ICA were reported in dose length product (DLP, milligray*cm) and dose area product (DAP, gray*cm2), respectively. DLP was converted to an effective dose (mSv) with a conversion factor of k = 0.014 and DAP with a conversion factor of k = 0.29. The effective doses were compare between patients who received both examinations.

Patients' symptoms were evaluated with the validated Seattle Angina Questionnaire 7 (SAQ7) via a single phone interview. Dyspnea was considered as an anginal symptom. All patients with SAQ7 Anginal Frequency score 100 were considered asymptomatic.

At the CTO PCI, optimal medical therapy was prescribed to all patients.

Stent- and patient-related characteristics examined in the study:

Age (years), body mass index (kg/m2), sex, smoking history, medical conditions at CTO PCI (diabetes, insulin required diabetes, heart failure, peripheral artery disease, dyslipidemia, hypertension, pulmonary disease, chronic kidney disease, atrial fibrillation, cardiac pacemaker, prior myocardial infarction, prior stroke, prior PCI, prior CABG), double-CTO (two treated CTO:s in one procedure), coronary artery dominance (RCA, left circumflex coronary artery (LCX), balanced)), a non-CTO stent implanted in the CTO PCI procedure, clinical presentation (stable angina pectoris or acute coronary syndrome), CCTA Agatston calcium score, stented vessel (RCA, left anterior descending artery (LAD), LCX), Japanese-CTO score (objective index of CTO procedure difficulty), long CTO stent parameters (number of consecutive stents, total stent length (mm), stent length in lesions stented with a single stent (mm), stent length in lesions stented with multiple stents (mm), stent diameter (mm)), duration of the follow-up since stent implantation (years).

The values are presented as medians and IQRs or n (%), as appropriate. The stent lengths are presented as medians and ranges (minimum-maximum).

Statistical analysis Descriptive statistics were reported with median and interquartile range (IQR) for continuous variables, and with frequency (%) for categorical variables. The demographic variables of the CCTA-positive group were compared to the corresponding variables of the CCTA-negative group. Categorical variables were analysed with Fisher's exact test or Pearson's chi-square test, and continuous or ordinal variables with Mann-Whitney U test. The alpha level was 0.05. CCTA performance in evaluating the patency of CTO stents was analysed with sensitivity, specificity, negative predictive value (NPV) and positive predictive value (PPV) in patients receiving both CCTA and ICA. ICA was the reference standard. All the statistical analyses were performed using SPSS version 28 (IBM).

ELIGIBILITY:
Inclusion Criteria:

* Surviving patients with a CTO PCI minimum of four years prior to the study date
* Successful CTO PCI with a drug-eluting stent
* Primary procedure minimum of four years prior to study date
* CTO stent length ≥ 38 mm in right coronary artery (RCA) and left anterior descending (LAD) coronary artery
* CTO stent length ≥ 30 mm in left circumflex coronary artery (LCX). The definition is clinical.
* Age at primary procedure ≤ 75 years
* Communication in English, Finnish or Swedish

Exclusion Criteria:

* Malignancy with poor prognosis or ongoing diagnostics
* Significantly impaired performance in daily activities
* Significant psychiatric disorder
* Active alcohol or drug abuse
* Memory disorder or other cognitive impairment
* Primary procedure in-stent CTO PCI
* Target vessel revascularisation or CABG after the primary - procedure
* Glomerular filtration rate ≤40 ml/min
* ICA or CCTA less than six months prior to the study date

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-01-16 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2024-06-08 (Actual)

PRIMARY OUTCOMES:
Stent patency assesment with third-generation dual-source CCTA | up to 7.3 months (maximum time between CCTA and ICA)
  Assessability of stent patency with third-generation dual-source CCTA in long coronary artery chronic total occlusion stents. CCTA results were divided into three categories: 1) negative (<50% stent luminal narrowing), 2) ISR (> 50% stent luminal narrowing) or 3) inconclusive (CCTA was not able to define the degree of stent luminal narrowing). Patients with ISR or inconclusive result were considered as CCTA positive. Confirmation imaging was conducted with ICA, if necessary. Positive predictive value, negative predictive value, sensitivity and specificity were calculated.

SECONDARY OUTCOMES:
To determine significant differences in distribution of patient- and lesion-related characteristics in third-generation dual-source CCTA negative versus positive patient groups. | through study completion, average of 1 year
  Patient-related characteristics assessed: age, body mass index, sex, smoking history, medical conditions at CTO PCI (diabetes, insulin required diabetes, heart failure, peripheral artery disease, dyslipidemia, hypertension, pulmonary disease, chronic kidney disease, atrial fibrillation, cardiac pacemaker, prior myocardial infarction, prior stroke, prior PCI, prior CABG), double-CTO (two treated CTO:s in one procedure), coronary artery dominance (RCA, LCX or balanced), a non-CTO stent implanted in the CTO PCI procedure, clinical presentation (stable or acute), CCTA Agatston calcium score.
  Lesion-related characteristics assessed: stented vessel (RCA, LAD, LCX), Japanese-CTO score (objective index of CTO procedure difficulty), long CTO stent parameters (number of consecutive stents, total stent length, stent length in lesions stented with a single stent, stent length in lesions stented with multiple stents, stent diameter), duration of the follow-up since stent implantation.
To compare radiation exposure of third-generation dual-source CCTA to ICA, measured as effective dose, in patients receiving both examinations. | from CCTA to possible ICA, up two 7.3 months
  Radiation exposure of third-generation dual-source CCTA (dose length product (DLP), milligray*cm) and radiation exposure of ICA (dose area product (DAP), gray*cm2) were converted to effective dose (millisievert, mSv) and compared.

CONTACTS AND LOCATIONS:
Overall Officials: Petri Laine, Ph.D., Principal Investigator — Department of Cardiology, Heart and Lung Center, Helsinki University Central Hospital
Locations (1):
- Helsinki University Central Hospital, Helsinki, Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: No